CLINICAL TRIAL: NCT04310189
Title: The Role of IL-22/IL-22BP Axis in Atopic Dermatitis. A Cross Sectional Monocentric Pilot Study
Brief Title: The Role of IL-22/IL-22BP Axis in Atopic Dermatitis
Acronym: DA/IL-22BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Plateforme CIMNA, Laboratoire d'Immunologie, Nantes University Hospital (Unknown); UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC19_0320
Record Dates: First submitted 2020-03-06; First posted 2020-03-17 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; eczema; interleukin 22
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biopsy — All patients will have a blood sample and 2 skin biopsies (2 mm diameter) in lesional and non lesional area

SUMMARY:
Interleukin 22 (IL-22) is known to be regulated by IL-22 binding protein (IL-22BP), a soluble, inhibitory receptor. The potential role of IL-22BP in atopic dermatitis (AD) is mostly unknown and deserves further investigation. The main objective of this study is to better understand the potential protective role of IL-22BP through the assessment of its expression at the Messenger Ribonucleic Acid (mRNA) and protein levels in skin and serum which will be correlated to the severity of the diseases and through the identification of its cellular sources in lesions. The results of this study will help to correctly interpret the levels of IL-22 in AD and will potentially allow identifying biomarkers for patient stratification and predicting clinical outcomes to targeted therapeutic agents.

DETAILED DESCRIPTION:
This is a single-visit study. All patients will have a blood sample and 2 skin biopsies (2 mm diameter) in lesional and non lesional area

. It is planned to include 45 patients (15 patients per severity group: SCORAD ]25-50] , ]50-65]; 50-65; >65).The first 20 patients included will be group 2 and 3 patients (SCORAD > 50).

The patients will be adults with AD recruited from the cohort of patients followed up in the Dermatology department of Nantes University Hospital. A refusal rate of 4/5 is expected. Recruitment can therefore be envisaged in 18 months (2.5 patients/month). Patients will be recruited during follow-up consultations or at the first consultation in the department. Recruitment will be coordinated by the clinical research team (CRT). Blood samples will be taken by the CRT Nurse. The skin and blood samples will be sent to the CIMNA/ Immunology Laboratory Nantes University hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients with AD according to UK Working Party criteria
* Patients affiliated to French social security system
* Patients who gave written consent after reading the protocol
* Moderate to severe AD (SCORAD score>25)
* Presence of at least one lesional and one non-lesional skin area in the area covered by the clothing
* No immunosuppressive systemic treatment in progress for at least 3 months or biologics for at least 4 months

Exclusion Criteria:

* Minor patients
* Pregnant and/or breastfeeding women
* Patients under guardianship or tutorship
* Inability to understand information and instructions
* Patients undergoing systemic immunosuppressive treatment for at least 3 months or biologics for at least 4 months
* Patient included in a clinical trial
* Documented allergy to the anesthetic (xylocain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Expression levels of IL-22 at the transcriptomic level | 1 day
  To compare the expression levels of IL-22 at the transcriptomic level in non lesional and lesional skin between the different groups of AD patients included in the study.
  Three groups of patients will be defined based on the SCORAD score . The score is out of 103 and is higher the greater the severity of the disease:
  * Group 1: SCORAD score between ]25-50]
  * Group 2: SCORAD between ]50; 65]
  * Group 3: SCORAD greater than 65.

SECONDARY OUTCOMES:
IL-22 expression levels in lesional skin at the protein level | 1 day
  To compare IL-22 expression levels in lesional skin at the protein level between the different AD patient groups included in the study.
expression levels of IL-22BP at the transcriptome level in in lesional skin | 1 day
  To compare the expression levels of IL-22BP at the transcriptome level in in lesional skin between the different groups of AD patients included in the study.
expression levels of IL-22BP at the protein level in lesional | 1 day
  To compare the expression levels of IL-22BP at the protein level in lesional skin between the different groups of AD patients included in the study.
level of IL22 gene expression in lesional and non lesional skin | 1 day
  To compare the level of IL22 gene expression in lesional and non lesional skin within each patient group
level of IL22BP gene expression in in lesional and non lesional | 1 day
  To compare the level of IL22BP gene expression in in lesional and non lesional in each patient group.
level of IL22R gene expression in lesional skin | 1 day
  To compare the level of IL22R gene expression in lesional skin between different groups of patients.
the level of IL22 receptor (IL22R ) gene expression in in lesional and non lesional skin | 1 day
  Compare the level of IL22 receptor (IL22R ) gene expression in in lesional and non lesional skin within each patient group
The level of expression of the following IL-22-induced genes | 1 day
  To compare the level of expression of the following IL-22-induced genes in injured skin between different groups of AD patients: S100A8, involucrin, loricrin
The level of IL-22-induced gene expression in lesional and non-lesional skin | 1 day
  To compare the level of IL-22-induced gene expression in lesional and non-lesional skin in each patient group: S100A8, involucrin, loricrin...
Level of IL-22BP and IL-22 proteins in serum | 1 day
  Measuring the level of IL-22BP and IL-22 proteins in serum
Locating IL-22 Binding protein (BP) | 1 day
  Locating IL-22 Binding protein (BP) producing cells in the lesional skin of patients with a SCORAD>50 (n = 10) (qualitative)
Characterizing IL-22 Binding protein (BP) | 1 day
  Characterizing (phenotype) IL-22 Binding protein (BP) producing cells in the lesional skin of patients with a SCORAD>50 (n = 10) (qualitative)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien BARBAROT, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided